CLINICAL TRIAL: NCT03570840
Title: Pediatric Metabolic Syndrome Study
Acronym: PMSS
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 19375; 0863 (Other: CTRC)
Record Dates: First submitted 2011-05-09; First posted 2018-06-27 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Metabolic Syndrome; Overweight and Obesity; Cardiovascular Risk Factor
Keywords: pediatric metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obese children and adolescents

SUMMARY:
The Pediatric Metabolic Syndrome Study is an observational study being conducted at the Medical University of South Carolina to investigate cardiometabolic risk parameters in obese subjects ages 4 to 21. A detailed assessment is performed on eligible subjects including fasting labwork, anthropometrics, nutrition analysis, body composition testing, echocardiography, and carotid IMT measurements.

ELIGIBILITY:
Inclusion Criteria:

age 4 to 21 years history of obesity (BMI at or over the 95th% for age/gender)

Exclusion Criteria:

age below 4 or above 21 years no history of obesity current pregnancy current chronic oral steroid use current insulin use

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: obese 4 to 21 yo subjects
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06-10 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
fasting insulin | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Melissa H Henshaw, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC, Charleston, South Carolina, United States